CLINICAL TRIAL: NCT04321980
Title: A Phase 1 Open-Label Single-Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of OP-101 (Dendrimer N-acetyl-cysteine) After Subcutaneous Administration in Healthy Volunteers
Brief Title: A Clinical Study to Measure the Effect of OP-101 After Being Administered Subcutaneous in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orpheris, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OP-101-003
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1 (Experimental): Subjects in Cohort 1 will be administered 4 mg/kg OP-101 as a subcutaneous (SC) injection.
  Interventions: Drug: OP-101
- Cohort 2 (Experimental): Subjects in Cohort 2 will be administered 8 mg/kg OP-101 as a SC injection.
  Interventions: Drug: OP-101

INTERVENTIONS:
Drug: OP-101 — Subcutaneous injection of OP-101 in healthy volunteers

SUMMARY:
A clinical study to measure the Safety, Tolerability, and Pharmacokinetics of OP-101 After Subcutaneous Administration in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Is a healthy man or woman age 18 to 65 years, inclusive, at the Screening Visit;
* Has the ability to understand and sign the written Informed Consent Form (ICF) and local medical privacy authorization forms, which must be obtained prior to any study related procedures being completed;
* Body mass index (BMI) between 18 and 32 kg/m2, inclusive;
* Is in general good health, based upon the results of a medical history assessment, physical examination, vital signs, and laboratory profile, as judged by the Investigator;
* Female subjects of non-childbearing potential must be either surgically sterile (hysterectomy, bilateral tubal ligation, salpingectomy, and/or bilateral oophorectomy at least 26 weeks before the Screening Visit) or postmenopausal, defined as spontaneous amenorrhea for at least 2 years, with follicle-stimulating hormone (FSH) in the postmenopausal range at screening, based on the central laboratory's ranges;
* Female subjects of childbearing potential (ie, ovulating, premenopausal, and not surgically sterile) and all male subjects must use a medically accepted contraceptive regimen (including hormonal contraceptives) during their participation in the study and for 30 days after the last administration of study drug. Medically accepted contraceptive methods are defined as those with 90% or greater efficacy;
* Acceptable methods of contraception for male subjects enrolled in the study include the following:

  • Condoms or surgical sterilization of subject at least 26 weeks before the Screening Visit (vasectomy);
* Acceptable methods of contraception for female subjects enrolled in the study include the following:

  * Surgical sterilization of subject at least 26 weeks before the Screening Visit (includes hysterectomy or bilateral tubal ligation, oophorectomy, or salpingectomy);
  * Intrauterine device for at least 12 weeks before the Screening Visit;
  * Hormonal contraception (oral, implant, injection, ring, or patch) for at least 12 weeks before the Screening Visit; or
  * Diaphragm;
* If male, subjects must agree to abstain from sperm donation through 90 days after administration of the last dose of study drug;
* Female subjects may not be pregnant, lactating, or breastfeeding;
* Female subjects of childbearing potential must have negative result for pregnancy test at screening and Check-in;
* Subjects must have a negative test result for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCVab), and human immunodeficiency virus (HIV) antibody at screening;
* Subjects must have an estimated glomerular filtration rate (eGFR) of ≥90 mL/min/1.73m2 at screening;
* Subjects must have a negative urine test for drugs of abuse (opiates, benzodiazepines, amphetamines, cannabinoids, cocaine, barbiturates, and phencyclidine), cotinine, and breath alcohol test at screening and Check-in; and
* Subjects must be willing and able to abide by all study requirements and restrictions.

Exclusion Criteria:

* Evidence of clinically significant hematologic, renal, endocrine, pulmonary, cardiac, gastrointestinal (GI), hepatic, psychiatric, neurologic, immunologic, allergic disease (including multiple or clinically significant drug allergies), or any other condition that, in the opinion of the Investigator, might significantly interfere with the absorption, distribution, metabolism, or excretion of study drug, or place the subject at an unacceptable risk as a participant in this study;
* History of malignancy (other than successfully treated basal cell or squamous cell skin cancer);
* History or presence of an abnormal ECG that, in the opinion of the Investigator, is clinically significant;
* Laboratory results (serum chemistry, hematology, coagulation, and urinalysis) outside the normal range at screening and Check-in and considered clinically significant in the opinion of the Investigator. Any elevation of aspartate transaminase (AST) and alanine transaminase (ALT) above the upper limit of normal at screening and/or Check-in is exclusionary. One retest of an exclusionary laboratory result is allowed at the discretion of the Investigator;
* Has had an acute illness considered clinically significant by the Investigator within 30 days prior to screening;
* History of alcoholism or drug abuse within 2 years prior to screening;
* Has used any product containing nicotine within 90 days prior to screening or intends to use any product containing nicotine during the course of the study;
* Has had any immunizations (live vaccines) in the 4 weeks prior to screening;
* Has used medications that affect GI motility or gastric emptying; such as metoclopramide, proton pump inhibitors, and H2 blockers; within 30 days prior to Day 1;
* Has used any prescription or over-the-counter medication (with exception of acetaminophen), vitamins/herbal supplements (with the exception of hormonal contraceptives) within 14 days prior to Day 1;
* Has used any other study drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to Day 1;
* Has lost or donated >450 mL of whole blood or blood products within 30 days prior to screening;
* Investigator has reason to believe that the subject may be unable to fulfill the protocol visit schedule or requirements;
* Has any finding that, in the view of the Investigator or Medical Monitor, would compromise the subject's safety requirements; or
* Is employed by the Sponsor, the Contract Research Organization (CRO), or the study site (permanent, temporary contract worker, or designee responsible for the conduct of the study), or is a family member (spouse, parent, sibling, or child) of the Sponsor, CRO, or study site employee.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 8 participants were enrolled and treated in the study.
Groups:
- Cohort 1: 4 mg/kg: Participants in Cohort 1 received a single dose of 4 milligram per kg (mg/kg) OP-101 as subcutaneous (SC) injection on Day 1.
- Cohort 2: 8 mg/kg: Participants in Cohort 2 received a single dose of 8 mg/kg OP-101 as SC injection on Day 1.
Period: Overall Study
Arm/Group | Cohort 1: 4 mg/kg | Cohort 2: 8 mg/kg
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety population which included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 4 mg/kg | Cohort 2: 8 mg/kg | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  White | 3 | 3 | 6
  Filipino | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. A TEAE (treatment-emergent adverse event) was defined as an AE that emerges, having been absent prior to the study, or an AE that worsens in severity after the first dose of the study drug. Serious AE (SAE) was an AE resulting in any of the following outcomes: death; life-threatening adverse event, required hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect, or a medically important event.
Time Frame: Up to Day 15
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: 4 mg/kg: Participants in Cohort 1 received a single dose of 4 mg/kg OP-101 as SC injection on Day 1.
Arm/Group | Cohort 1: 4 mg/kg | Cohort 2: 8 mg/kg
Number analyzed (Participants) | 4 | 4
Participants
  Any TEAE | 2 | 3
  Any SAE | 0 | 0

2. Secondary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax) of OP-101
Description: Cmax: maximum observed plasma concentration.
Time Frame: Pre-dose, 0.5 hours and 1, 2, 4, 6, 8, 10, 12, 16, 24, 30-36, 48 hours post-dose
Population: Analysis was performed on pharmacokinetic (PK) parameter population which was defined as all participants who received a dose of study drug and had at least 1 PK parameter.
Measure: Mean (Standard Deviation); unit: microgram per milliliter(mcg/mL)
Arm/Group | Cohort 1: 4 mg/kg | Cohort 2: 8 mg/kg
Number analyzed (Participants) | 4 | 4
microgram per milliliter(mcg/mL) | 3.473 (0.8183) | 6.640 (0.6073)

3. Secondary Outcome: Pharmacokinetics: Time to Reach Maximum Plasma Concentration (Tmax) of OP-101
Description: Tmax: time to reach maximum observed plasma concentration.
Time Frame: Pre-dose, 0.5 hours and at 1, 2, 4, 6, 8, 10, 12, 16, 24, 30-36, 48 hours post-dose
Population: Analysis was performed on PK parameter population.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: 4 mg/kg | Cohort 2: 8 mg/kg
Number analyzed (Participants) | 4 | 4
hours | 14.015 [10.00 to 16.05] | 16.000 [12.00 to 24.05]

4. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-last) of OP-101
Description: AUC0-last: Area under the concentration versus time curve from time zero to the last quantifiable concentration (Clast).
Time Frame: Pre-dose, 0.5 hours and 1, 2, 4, 6, 8, 10, 12, 16, 24, 30-36, 48 hours post-dose
Population: Analysis was performed on PK parameter population.
Measure: Mean (Standard Deviation); unit: hr*mcg/mL
Arm/Group | Cohort 1: 4 mg/kg | Cohort 2: 8 mg/kg
Number analyzed (Participants) | 4 | 4
hr*mcg/mL | 80.940 (51.8190) | 212.325 (30.6459)

5. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time Zero to 48 Hour Post Dose Time Point (AUC0-48) of OP-101
Description: Area under the concentration versus time curve from time zero to 48 hour post dose time point.
Time Frame: Pre-dose, 0.5 hours and 1, 2, 4, 6, 8, 10, 12, 16, 24, 30-36, 48 hours post-dose
Population: Analysis was performed on PK parameter population.
Measure: Mean (Standard Deviation); unit: hr*mcg/mL
Arm/Group | Cohort 1: 4 mg/kg | Cohort 2: 8 mg/kg
Number analyzed (Participants) | 4 | 4
hr*mcg/mL | 121.705 (16.9069) | 222.173 (12.4690)

6. Secondary Outcome: Pharmacokinetics: Renal Clearance (CLR) for OP-101
Description: CLR was defined as renal clearance of the drug from plasma utilizing the AUC and cumulative amount of unchanged study drug excreted into the urine (Ae) to the same duration (as Amount recovered/AUC at 0-48 hours).
Time Frame: Pre-dose, 0 to 4, 4 to 8, 8 to 12, 12 to 18, 18 to 24, and 24 to 48 hours post dose
Population: Analysis was performed on PK parameter population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: liter per hour (L/hr)
Arm/Group | Cohort 1: 4 mg/kg | Cohort 2: 8 mg/kg
Number analyzed (Participants) | 2 | 4
liter per hour (L/hr) | 0.175 (0.0354) | 0.150 (0.0606)

ADVERSE EVENTS:
Time Frame: Up to Day 15
Description: Analysis was performed on safety population.
Arm/Group | Cohort 1: 4 mg/kg | Cohort 2: 8 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/4 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 4 mg/kg (N=4) | Cohort 2: 8 mg/kg (N=4)
Injection site erythema (General disorders) | 0 | 3
Injection site mass (General disorders) | 0 | 1
Injection site pain (General disorders) | 1 | 0
Injection site pallor (General disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT04321980/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT04321980/SAP_001.pdf